CLINICAL TRIAL: NCT00375167
Title: Efficacy of the Recovery Workbook as a Psychoeducational Tool for Facilitating Recovery in Persons With Severe and Persistent Mental Illness
Brief Title: Efficacy of the Recovery Workbook as a Psychoeducational Tool for Facilitating Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Terry Krupa, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2018-11

CONDITIONS: Mental Disorders
Keywords: Recovery, Hope, Empowerment, Randomized Control Trial
MeSH Terms: conditions — Mental Disorders; Empowerment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recovery Workbook Intervention (Experimental): 12-week Recovery Intervention: The intervention is a 12-week group-based intervention. The intervention is informed by the Recovery Workbook- a validated intervention for people with serious mental illness. The intervention includes 2 hour sessions for 12 weeks that focus on the following areas: Introduction to the intervention; Recovery; Knowledge and Control; Managing life stress; Enhancing personal meaning; Building personal support; and Setting personal goals. The total time period of the intervention is 24 hours. Participants in this arm also receive treatment as usual.
  Interventions: Behavioral: Recovery Workbook Training (psychoeducational training); Behavioral: ACT as usual
- Treatment as usual (No Intervention): The participants in the control arm will continue to receive treatment as usual. TAU is Assertive Community Treatment. Assertive Community Treatments are structured to meet set fidelity standards that are evidence-based. This arm did not receive any intervention.

INTERVENTIONS:
Behavioral: Recovery Workbook Training (psychoeducational training) — The Recovery Workbook uses an educational process to increase awareness of recovery, increase knowledge and control of the illness, increase awareness of the importance and nature of stress, enhance personal meaning, build personal support, and develop goals and plans of action. The intervention period of 30 weekly sessions recommended by Spaniol and colleagues was shortened to 12 weekly sessions to accommodate for clinical and participant commitment. No workbook content was excluded, and all practice exercises were covered.
  Arms: Recovery Workbook Intervention
Behavioral: ACT as usual — Assertive Community Treatment services provided as per established and evidence-based fidelity standards.
  Arms: Recovery Workbook Intervention

SUMMARY:
The present study will determine if Spaniol and colleague's (1994) Recovery Workbook group intervention is an effective clinical tool to move a person with SMI along in their journey of recovery. The primary outcome measurements of this study will be the participants' perceived level of empowerment, hope and optimism, knowledge of recovery, and life satisfaction. This kind of information would add to the current body of knowledge about how principles of recovery can be used in psychoeducational programs used by outpatient community mental health services.

DETAILED DESCRIPTION:
ABSTRACT:

Objective: Adopting the principles of recovery into the mental health field has been a growing area for discussion at many different levels of care. The present study will determine if Spaniol and colleague's (1994) Recovery Workbook group intervention can be used as an effective clinical tool to move a person with a severe mental illness along in their journey of recovery. The primary outcome measurements of this study will be the participants' perceived level of empowerment, hope and optimism, knowledge of recovery, and life satisfaction. Method: The study will be a multicenter, prospective, single-blinded, randomized control trial. Sixty participants will be recruited from three Assertive Community Treatment Teams (ACTT) in Kingston, Ontario and individuals will be randomized to either the control or intervention arm of the study. The control arm of the study will receive their regular services from ACTT. The intervention arm will participate in a 10-week psychoeducational group program in addition to receiving their regular services from ACTT. Results: Analysis will be performed by intention to treat, based on total scores of four assessments which will be performed at the trial commencement and termination.

ELIGIBILITY:
Inclusion Criteria:

1. Receive support from an Assertive Community Treatment Team.
2. Meet the DSM-IV diagnostic classification for schizophrenia, schizoaffective, schizophreniform, delusional disorder, or bipolar disorder.
3. Aged 18-55 years-old.
4. Individuals agree to participate in the study after they have been informed of all the expected benefits and risks.
5. Neither substance misuse nor organic disorder judged to be the major cause of psychotic symptoms.

Exclusion Criteria:

1. Inability to give informed consent
2. Diagnosis of dementia
3. Significant head injury or other brain injury leading to cognitive impairment
4. Mental retardation (premorbid IQ < 65)
5. Require an interpreter

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-09; Primary Completion 2007-01 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Skye Barbic, BScOT, Principal Investigator — Queen's University; Terry Krupa, PhD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Managers of 2 ACT teams reviewed all clients to identify those eligible for study between August and October 2006. Eighty-one identified and informed about the study, with 34 people providing informed consent. Clients were grouped by team and then randomized to one of the two arms. One person dropped out at time of randomization
Pre-assignment Details: Participants were grouped according to team prior to randomization because the group intervention was administered by team
Groups:
- ACT With Recovery Workbook: Recovery Workbook (Psychoeducation training) Clients of Assertive Community Treatment randomized to condition receiving the Recovery Workbook intervention in a group format over 12 weeks. The sessions focus on the following areas: Introduction; Recovery; Knowledge and Control; Managing life stress; Enhancing personal meaning; Building personal support and; Setting personal goals
  Recovery Workbook Training (psychoeducational training): The Recovery Workbook uses an educational process to increase awareness of recovery, increase knowledge and control of the illness, increase awareness of the importance and nature of stress, enhance personal meaning, build personal support, and develop goals and plans of action. The intervention period of 30 weekly sessions recommended by Spaniol and colleagues was shortened to 12 weekly sessions to accommodate for clinical and participant commitment. No workbook content was excluded, and all practice exercises were covered.
- ACT as Usual: Assertive community Treatment The participants were clients of Assertive Community Treatment receiving standard treatment as usual. Assertive Community Treatments are structured to meet set fidelity standards that are evidence-based.
  ACT as usual: Assertive Community Treatment services provided as per established and evidence-based fidelity standards.
Period: Overall Study
Arm/Group | ACT With Recovery Workbook | ACT as Usual
Started | 16 (Clients were already receiving ACT services and this continued after study completion) | 17 (Participants were already clients of ACT and continued receiving services following this period)
Completed | 16 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All statistical analyses were intent-to-treat analyses. Demographic differences between the teams and between the intervention and control groups were analyzed by using t tests and chi square tests.
Groups:
- Total: Total of all reporting groups
Arm/Group | ACT With Recovery Workbook | ACT as Usual | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 44.69 (9.62) | 44.58 (8.05) | 44.62 (8.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 11 | 11 | 22
Hope, Empowerment, Recovery, QOL [Mean (Standard Deviation); unit: units on a scale]
  Hope | 37.13 (6.53) | 36.00 (5.36) | 36.54 (5.38)
  Empowermeent | 61.96 (6.91) | 63.88 (6.91) | 62.95 (6.87)
  Quality of Life | 20.34 (5.01) | 20.70 (4.13) | 20.53 (4.51)
  Recovery | 163.75 (22.60) | 156.41 (14.22) | 159.97 (18.87)

OUTCOME MEASURES:

1. Primary Outcome: Hope Herth Index
Description: The Herth Hope Index was used to gather information about participants' level of hopefulness. The 12-item scale is easily administered and has been used with persons with serious mental illness . It is a self-report tool, and respondents answer on a 4-point agreement scale that ranges from "strongly disagree" to "strongly agree". The scoring range is from 12-48 with a higher score indicating higher levels of hope. The scale has been shown to have an alpha coefficient of .97 and a test-retest reliability of .91 within two weeks. Criterion-related validity has also been supported by high correlations (.81-.92) with instruments measuring the same construct.
Time Frame: Within 3 days of completion of intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ACT With Recovery Workbook: Recovery Workbook These participants were clients of Assertive Community Treatment who were randomized to condition where in addition to usual service they received the Recovery Workbook intervention in a group format over 12 weeks. The sessions focus on the following areas: Introduction; Recovery; Knowledge and Control; Managing life stress; Enhancing personal meaning; Building personal support and; Setting personal goals
  Recovery Workbook Training:The Recovery Workbook uses an educational process to increase awareness of recovery, increase knowledge and control of the illness, increase awareness of the importance and nature of stress, enhance personal meaning, build personal support, and develop goals and plans of action. The intervention period of 30 weekly sessions recommended by Spaniol and colleagues was shortened to 12 weekly sessions to accommodate for clinical and participant commitment. No workbook content was excluded, and all practice exercises were covered.
Arm/Group | ACT With Recovery Workbook | ACT as Usual
Number analyzed (Participants) | 16 | 17
units on a scale | 38.93 (5.34) | 35.06 (5.36)

2. Primary Outcome: Empowerment Scale
Description: The construct measured is empowerment. The Empowerment Scale is a self-reported measure that contains 28 statements about empowerment to which participants respond on a 4-point agreement scale. Scoring range is 28-112, with a lower score indicating higher empowerment. Studies have demonstrated the scale's high internal consistency ({alpha}=.85-.90) and good reliability ({alpha}>.60) and validity (28,31,32).
Time Frame: Within 3 days of completion of interventions
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ACT With Recovery Workbook: Recovery Workbook These participants were clients of Assertive Community Treatment who were randomized to condition where in addition to usual service they received the Recovery Workbook intervention in a group format over 12 weeks. The sessions focus on the following areas: Introduction; Recovery; Knowledge and Control; Managing life stress; Enhancing personal meaning; Building personal support and; Setting personal goals
  Recovery Workbook Training: The Recovery Workbook uses an educational process to increase awareness of recovery, increase knowledge and control of the illness, increase awareness of the importance and nature of stress, enhance personal meaning, build personal support, and develop goals and plans of action. The intervention period of 30 weekly sessions recommended by Spaniol and colleagues was shortened to 12 weekly sessions to accommodate for clinical and participant commitment. No workbook content was excluded, and all practice exercises were covered.
Arm/Group | ACT With Recovery Workbook | ACT as Usual
Number analyzed (Participants) | 16 | 17
units on a scale | 55.93 (6.91) | 61.96 (7.33)

3. Primary Outcome: Recovery Assessment Scale
Description: The construct is Personal Recovery, defined as a person's ability to live a full and meaningful life. The Recovery Assessment Scale (RAS) has 41-items and uses a 5-point agreement scale, and a total score is used, with scores ranging from 41-205, with a higher score indicating a higher sense of personal recovery. The RAS also has 5 subscales (see below). Subscales are added to produce a total score. Domain 1 is Confidence and Hope. he scoring range here is 9-45, where a higher score indicating higher recovery. Domain 2 is Willingness to Ask for Help. Scoring range is 3-15. Domain 3: Ability rely on others: Scoring range 5-25. Domain 4 Symptoms: Scoring range 4-20. Domain 5: Goal and Success Orientation: Scoring range 3-15. For each domain, higher values represent a better outcome.
Time Frame: Within 3 days of completion of intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ACT With Recovery Workbook: Recovery Workbook : These participants were clients of Assertive Community Treatment who were randomized to condition where in addition to usual service they received the Recovery Workbook intervention in a group format over 12 weeks. The sessions focus on the following areas: Introduction; Recovery; Knowledge and Control; Managing life stress; Enhancing personal meaning; Building personal support and; Setting personal goals
  Recovery Workbook Training: The Recovery Workbook uses an educational process to increase awareness of recovery, increase knowledge and control of the illness, increase awareness of the importance and nature of stress, enhance personal meaning, build personal support, and develop goals and plans of action.The intervention period of 30 weekly sessions recommended by Spaniol and colleagues was shortened to 12 weekly sessions to accommodate for clinical and participant commitment. No workbook content was xcluded, and all practice exercises were covered.
Arm/Group | ACT With Recovery Workbook | ACT as Usual
Number analyzed (Participants) | 16 | 17
units on a scale
  Recovery total | 168.81 (20.11) | 149.11 (22.09)
  Confidence and Hope | 37.13 (5.51) | 31.82 (7.92)
  Willingness to Ask for Help | 12.00 (2.33) | 11.11 (1.73)
  Ability rely on others | 21.31 (2.91) | 18.35 (4.74)
  Symptoms | 17.18 (1.79) | 14.76 (2.61)
  Goal and Success Orientation | 11.75 (2.11) | 9.65 (2.62)

4. Primary Outcome: Quality of Life Index, General Version
Description: The Quality of Life Index, General Version (37), is a 33-item self-report scale measuring satisfaction with and importance of aspects of life. It includes four subscales: health and functioning, socioeconomic status, psychological status, and significant others. Satisfaction and importance are measured on a 6-point agreement scale. A high score indicates higher quality of life. Full scoring instructions and computer algorithm is available at http://qli.org.uic.edu/questionaires/pdf/genericversionIII/genericscoring.pdf. Importance ratings are used to weight satisfaction responses so that scores reflect satisfaction with aspects of life that are valued by the individual (37). For internal consistency and reliability, Cronbach's alpha is .92 for the entire tool and .88, .75, .80, and .68, respectively, for the subscales (37). Possible range for the final scores = 0 to 30, where a higher value represents a better outcome..
Time Frame: Within 3 days of completion of intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACT With Recovery Workbook | ACT as Usual
Number analyzed (Participants) | 16 | 17
units on a scale | 20.34 (5.01) | 20.70 (4.13)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | ACT With Recovery Workbook | ACT as Usual
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No